CLINICAL TRIAL: NCT03252951
Title: An Innovative Rehabilitation Approach for Women With Anal Incontinence
Brief Title: Physical Therapy for Anal Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Lori Tuttle, Associate Professor, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 141728
Record Dates: First submitted 2017-08-14; First posted 2017-08-17 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Anal Incontinence; Fecal Incontinence
MeSH Terms: conditions — Encopresis; Fecal Incontinence | interventions — Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Eccentric Training (Experimental)
  Interventions: Behavioral: Eccentric Training
- Concentric Training (Experimental)
  Interventions: Behavioral: Concentric Training
- Isometric Training (Experimental)
  Interventions: Behavioral: Isometric Training
- Biofeedback (Active Comparator)
  Interventions: Behavioral: Biofeedback

INTERVENTIONS:
Behavioral: Eccentric Training — Different Anal Sphincter Exercise Types for muscle hypertrophy
  Arms: Eccentric Training
Behavioral: Concentric Training — Different Anal Sphincter Exercise Types for muscle hypertrophy
  Arms: Concentric Training
Behavioral: Isometric Training — Different Anal Sphincter Exercise Types for muscle hypertrophy
  Arms: Isometric Training
Behavioral: Biofeedback — Standard of Care Biofeedback Training
  Arms: Biofeedback

SUMMARY:
Anal incontinence is a significant public health problem estimated to affect 7-15% of women in the United States. Traditional rehabilitation strategies include biofeedback and Kegel exercises for pelvic floor muscle strengthening, but this strategy does not incorporate strategies for resistance training that are known to cause muscle strengthening and hypertrophy in other muscles in the body. This study aims to investigate whether a novel pelvic floor resistance exercise program will increase pelvic floor muscle strength and improve anal incontinence and has the potential to impact rehabilitation strategies for the millions of women affected anal incontinence.

DETAILED DESCRIPTION:
The current proposal is focused on examining whether a novel resistance exercise program for the pelvic floor will strengthen pelvic floor muscles and improve symptoms in women with anal incontinence. Anal incontinence is a significant public health issue that is estimated to impact 7-15% of women. Traditional rehabilitation strategies such as Kegel exercises and biofeedback are a noninvasive strategy designed to strengthen the pelvic floor muscles, however, these exercises are performed with no resistance. There is a large body of evidence indicating that for muscle strengthening and hypertrophy to occur, exercises must be performed against resistance. Therefore, we have designed a novel exercise program for the pelvic floor that incorporates principals of resistance training known to be effective in other muscles in the body. The long-term goal of this research is to determine the most appropriate noninvasive strategies and interventions to improve pelvic floor function and symptoms of anal incontinence. This project is the first step in achieving this goal. The overall purpose of the current proposal is to determine whether novel physical therapy interventions are more effective than traditional biofeedback strategies in the treatment of anal incontinence. The specific aims of the proposal are: (1) To describe the use of the Functional Lumen Imaging Probe (FLIP) for pelvic floor exercise; (2) To determine whether eccentric, concentric, or isometric exercise training of the pelvic floor has a positive impact on the pelvic floor muscles and on symptoms of anal incontinence compared to traditional biofeedback training; (3) To determine whether using the FLIP in the vagina is as effective as its use in the anal canal for treatment of anal incontinence. To test these aims, the approach includes a randomized controlled exercise trial with use of validated measures of muscle function, muscle hypertrophy and validated symptom measures. This proposal describes an innovative approach to rehabilitation of the pelvic floor muscles that will provide information about pelvic floor function and that has the potential to shift the treatment paradigm for women with pelvic floor disorders.

ELIGIBILITY:
Inclusion Criteria:

* AI based on FISI questionnaire
* FISI scores between 10 and 45
* able to voluntarily contract pelvic floor muscles based on manometry measures

Exclusion Criteria:

* FISI score below 10 (mild disease) or greater than 45 (severe disease)
* manometry measure below the 10th percentile of normal (lack of muscle) or above 70th percentile of normal (little room to improve strength)
* history of large external hemorrhoids or history of bleeding hemorrhoids; co-existing inflammatory bowel disease
* constipation that is directly linked to neurological conditions such as spinal and peripheral nerve pathologies
* large pelvic organ prolapse (greater than stage 3)
* inability to contract the pelvic floor muscles on command
* pregnancy

Min Age: 22 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Length Tension Manometry after 12 weeks | 12 weeks
  change from baseline to 12 weeks

SECONDARY OUTCOMES:
Change in Muscle Hypertrophy (Ultrasound) after 12 weeks | 12 weeks
  change from baseline to 12 weeks
Change in FISI score after 12 weeks | 12 weeks
  change from baseline to 12 weeks

OTHER OUTCOMES:
Change in Length Tension Manometry after 1 year | 12 months
  change from baseline to 12 months
Change in Length Tension Manometry after 2 years | 24 months
  change from baseline to 24 months
Change in Muscle Hypertrophy (ultrasound) after 1 year | 12 months
  change from baseline to 12 months
Change in Muscle Hypertrophy (ultrasound) after 2 years | 24 months
  change from baseline to 24 months
Change in FISI score after 1 year | 12 months
  change from baseline to 12 months
Change in FISI score after 2 years | 24 months
  change from baseline to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Lori Tuttle, PT, PhD, Principal Investigator — San Diego State University
Locations (1):
- University of California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No